CLINICAL TRIAL: NCT00084214
Title: A Two-Stage Trial of STA-4783 in Combination With Weekly Paclitaxel for Treatment of Patients With Metastatic Melanoma
Brief Title: STA-4783/Paclitaxel or Paclitaxel Alone in Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4783-03
Record Dates: First submitted 2004-06-09; First posted 2004-06-10 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2008-12

CONDITIONS: Melanoma
Keywords: metastatic; increased antitumor effect
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — elesclomol; Paclitaxel

INTERVENTIONS:
Drug: STA-4783
Drug: Paclitaxel

SUMMARY:
This study is designed to assess the efficacy of a weekly treatment regimen of STA-4783 and paclitaxel in comparison to paclitaxel alone on tumor response in metastatic melanoma patients.

DETAILED DESCRIPTION:
STA-4783 is a taxane potentiator, enhancing the effect of antitumor response of paclitaxel. In an attempt to improve efficacy, paclitaxel is sometimes used in combination with other anticancer agents. When paclitaxel is combined with other anticancer agents, although response rate is usually increased, side effects are usually increased as well. There is an urgent need for agents that can enhance the antitumor effects of paclitaxel without further increasing undesirable side effects.

ELIGIBILITY:
Inclusion Criteria:

* M or F 18 or older with histologically confirmed metastatic (Stage IV) melanoma of cutaneous origin
* ECOG performance status of greater than or equal to 2
* Measurable disease per RECIST criteria
* Received no more than 1 regimen of prior chemotherapy (unlimited immunotherapy regimens are allowed)
* At least 4 weeks have passed since last chemotherapy or immunotherapy
* At least 2 weeks have passed since last radiotherapy.
* Life expectancy of greater than 12 weeks
* Clinical lab values within protocol parameters

Exclusion Criteria:

* Female patients pregnant or lactating
* Female patients of childbearing potential not using or not willing to use effective contraception
* Presence of a second malignancy other than nonmelanoma skin cancer
* Presence of a clinically significant and uncontrolled infection
* Presence of clinically significant arrythmias
* Presence of serious concurrent illness or other conditions that do not permit adequate follow-up and compliance with protocol
* History of severe hypersensitivity reactions to taxanes
* Use of any investigational agents within 4 weeks prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103
Dates: Start 2004-05

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Univ Of Arkansas/Arkansas Research Center, Little Rock, Arkansas
  - Scripps Cancer Center, San Diego, California
  - Northern California Melanoma Center, San Francisco, California
  - Cancer Institute Medical Group, Inc, Santa Monica, California
  - Anschutz Cancer Pavillion - Univ Of Colorado, Aurora, Colorado
  - Hematology Oncology P.C., Stamford, Connecticut
  - Medical Oncology and Hematology, P.C., Waterbury, Connecticut
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Research Institute Hawaii Pacific Health, Honolulu, Hawaii
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Oncology Specialists, Park Ridge, Illinois
  - Cancer Care Center Of Southern Indiana, Bloomington, Indiana
  - Center For Cancer Care At Goshen Health, Goshen, Indiana
  - Indiana Oncology Hematology Consultants, Iindianapolis, Indiana
  - Cancer Care Center, New Albany, Indiana
  - James Graham Brown Cancer Center - University Of Louisville, Louisville, Kentucky
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Ellis Fischels Cancer Center - Univ Of Missouri, Columbia, Missouri
  - Mountainside Hospital, Suburban Surgical Associates, St Louis, Missouri
  - Piedmont Oncology Specialists, Charlotte, North Carolina
  - Odyssey Research and St. Alexius Medical Center, Bismarck, North Dakota
  - Providence Cancer Center, Portland, Oregon
  - Danville Hematology & Oncology, Inc., Danville, Virginia
  - Office of James Stark, MD, Portsmouth, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - University of Wisconsin Medical School, Madison, Wisconsin